CLINICAL TRIAL: NCT06832020
Title: Avaliação Do Desenvolvimento Adaptativo a Longo Prazo Após a Cirurgia De Epilepsia Em Crianças E Adolescentes Farmacorresistentes
Brief Title: Determinants of Adaptive Behavior Through the Vineland Scale in Pediatric Patients with Severe and Drug-resistant Epilepsy
Status: Completed | Type: Observational
Sponsor: Ana Valeria Duarte Oliveira (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor-Investigator, Ana Valeria Duarte Oliveira, Doctor of Neurology, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 4.829.087
Record Dates: First submitted 2024-12-19; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy (treatment Refractory)
Keywords: Epilepsy Drug-resistant. Epilepsy Surgery. Vineland. Pediatrics patients
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Control group consisting of 204 patients and clinical group comprising 165 patients.: The patients were divided into two groups: a control group consisting of 204 patients without an established epileptogenic focus, and a clinical group comprising 165 patients with a diagnosed epilepsy, both groups, treated at the Ribeirão Preto Epilepsy Surgery Program (CIREP) of the Clinical Hospital of Ribeirão Preto - University of São Paulo (HCFMRP-USP) between 1996 and 2019.

SUMMARY:
Our interest in studying how pediatric patients develop after epilepsy surgery stems from the fact that difficult-to-control epilepsy causes changes in the brain's formation or functioning, leading some patients to experience slower development compared to others. By gaining a better understanding of how pediatrics patients fare after epilepsy surgery, specifically regarding their independence in daily activities (such as bathing or making the bed), their relationships with family and friends, their mobility, and their speech (whether it is understandable) we can learn more about patient recovery. The goal of this research is to determine whether, 4 years after epilepsy surgery, pediatrics patients show improvements in development. This study is important because it investigates what happens to the development of children who have undergone epilepsy surgery after a long period has passed since the procedure. Research focusing on long-term post-surgical outcomes is necessary, especially in pediatrics, as a brain is not fully developed and requires time to recover after surgery.

DETAILED DESCRIPTION:
Participation in the study was voluntary, and refusal to participate or withdrawal of consent at any of the three phases of the research did not result in any penalties. We are committed to maintaining the confidentiality of your child's data, and they were not identified. The data related to the clinical information for the purposes of this research were processed and stored in a database at the Epilepsy Surgery Center (CIREP) of the Hospital das Clínicas de Ribeirão Preto, where only the researchers had access via password. These data will be used for research purposes to assist in the planning of therapeutic intervention.

Once the inclusion in this study was identified and confirmed, the data of all patients were analyzed through a review of electronic medical records and the SAME (Medical and Statistical Archive Service) of HCFMRP-USP. The information obtained was stored in an SPSS database and subsequently analyzed. The following variables were collected: sex, age, age at pre- and postoperative neuropsychological assessment, Engel classification, type of surgery, resection, pathology, seizure frequency, dates of assessments, MRI reports, and findings from the Vineland scale related to communication, socialization, daily living skills, motor skills, and conclusions. Only the principal investigator was authorized to handle the database, in accordance with the data protection and confidentiality standards for the information collected from the patients' electronic medical records included in the study.

This study was classified as an observational retrospective cohort analysis. A total of 369 patients with chronological age ranging from 0 to 18 years and severe epilepsy that was unresponsive to drug therapy (defined as uncontrolled epilepsy despite the use of one or two combined drugs) were referred to the study. The patients were divided into two groups: a control group consisting of 204 patients without an established epileptogenic focus, and a clinical group comprising 165 patients with a diagnosed epilepsy, both groups, treated at the Ribeirão Preto Epilepsy Surgery Program (CIREP) of the Clinical Hospital of Ribeirão Preto - University of São Paulo (HCFMRP-USP) between 1996 and 2019.

The statistical analyses were conducted using the IBM SPSS 23.0 for Windows software (Statistical Package for Social Sciences, SPSS Inc., 1989-2004, Chicago, IL, USA). The variables were assessed for normality using the Kolmogorov-Smirnov test. Categorical variables were summarized using frequency counts, relative frequencies, and valid percentages. Continuous variables were presented as means and standard deviations, along with minimum and maximum values, median, and interquartile range. Univariate analysis was undertaken using post hoc Tukey to examine potential etiological differences between-subjects. Statistical analyses were performed using Pearson's correlation test, and multiple linear regression were conducted to identify neurologic predictors of adaptive function. A significance level of 0.05 or less was considered as the threshold for statistical significance.

The sample size was calculated using the G*Power 3.1.9.7 for Windows program (2020). We used Fisher's exact test, where the test power was set to 0.8, and the error probability was set to 0.05, indicating that the ideal total sample size would be 88 patients, distributed in two equally sized groups. We chose to conduct the study with all patients in the CIREP database, resulting in a sample composed of 369 pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age ranging from 0 to 18 years
* Severe epilepsy that was unresponsive to drug therapy (defined as uncontrolled epilepsy despite the use of one or two combined drugs) were referred to the study.

Exclusion Criteria:

* Involved patients whose parents or responsible relatives had psychiatric disorders
* Patients who were unable to complete the neuropsychological assessment questionnaire.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study was classified as an observational retrospective cohort analysis. A total of 369 patients with chronological age ranging from 0 to 18 years and severe epilepsy that was unresponsive to drug therapy (defined as uncontrolled epilepsy despite the use of one or two combined drugs) were referred to the study. The patients were divided into two groups: a control group consisting of 204 patients without an established epileptogenic focus, and a clinical group comprising 165 patients with a diagnosed epilepsy, both groups, treated at the Ribeirão Preto Epilepsy Surgery Program (CIREP) of the Clinical Hospital of Ribeirão Preto - University of São Paulo (HCFMRP-USP) between 1996 and 2019.
Sampling Method: Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Determinants of Changes in Adaptive Scores through the Vineland Scale in Pediatric Patients with Drug-Resistant Epilepsy | "From enrollment to the end of treatment at 48 months"
Determinants of Changes in Adaptive Scores through the Vineland Scale in Pediatric Patients with Drug-Resistant Epilepsy | "From enrollment to the end of treatment at 48 months"
  In a retrospective study, our objective was to assess the clinical condition of the patients through data such as Vineland Adaptive Behavior Scales (VABS) in pediatric patients with severe, difficult-to-control epilepsy. The VABS assesses various domains, including communication, daily living skills, socialization, and motor skills. The assessments were conducted in a blinded manner to avoid contaminating the data collection and results with any information obtained prior to the completion of the questionnaire.
  Regarding the performance of a given activity, a score of 2 indicates "yes, normally," 1 "sometimes or partially," and 0 "no, never." The 'N' scores indicate that the individual "has no opportunity" to perform the activity, and 'D' indicates "unknown," meaning the caregiver or responsible person does not know whether the patient performs the activity. The higher the score, the better the adaptive outcome the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tonicarlo R Velasco, Doctor, Study Director — Center for Pediatric Epilepsy Surgery, University Hospital, Ribeirão Preto Medical School, University of São Paulo, Brazil.
Locations (1):
- Center for Pediatric Epilepsy Surgery, University Hospital, Ribeirão Preto Medical School, University of São Paulo, Brazil., Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
A description of the complete protocol study will be provided so that the fases can be fully interpreted.
Supporting Information: Study Protocol
Time Frame: Beginning December 2025 and ending 2 years after the publication of results.
Access Criteria: The data related to this article will be available for public access through a link to the chosen academic journal.

REFERENCES:
- [Background] Vendrame M, Alexopoulos AV, Boyer K, Gregas M, Haut J, Lineweaver T, Wyllie E, Loddenkemper T. Longer duration of epilepsy and earlier age at epilepsy onset correlate with impaired cognitive development in infancy. Epilepsy Behav. 2009 Nov;16(3):431-5. doi: 10.1016/j.yebeh.2009.08.008. Epub 2009 Sep 19. PMID 19767243
- [Background] Nolan MA, Redoblado MA, Lah S, Sabaz M, Lawson JA, Cunningham AM, Bleasel AF, Bye AM. Intelligence in childhood epilepsy syndromes. Epilepsy Res. 2003 Feb;53(1-2):139-50. doi: 10.1016/s0920-1211(02)00261-9. PMID 12576175
- [Background] Loring DW, Meador KJ. Cognitive side effects of antiepileptic drugs in children. Neurology. 2004 Mar 23;62(6):872-7. doi: 10.1212/01.wnl.0000115653.82763.07. PMID 15037684
- [Background] Pulsifer MB, Brandt J, Salorio CF, Vining EP, Carson BS, Freeman JM. The cognitive outcome of hemispherectomy in 71 children. Epilepsia. 2004 Mar;45(3):243-54. doi: 10.1111/j.0013-9580.2004.15303.x. PMID 15009226
- [Background] Howell KB, Harvey AS, Archer JS. Epileptic encephalopathy: Use and misuse of a clinically and conceptually important concept. Epilepsia. 2016 Mar;57(3):343-7. doi: 10.1111/epi.13306. Epub 2016 Jan 18. PMID 26778176
- [Background] Fisher RS, Cross JH, D'Souza C, French JA, Haut SR, Higurashi N, Hirsch E, Jansen FE, Lagae L, Moshe SL, Peltola J, Roulet Perez E, Scheffer IE, Schulze-Bonhage A, Somerville E, Sperling M, Yacubian EM, Zuberi SM. Instruction manual for the ILAE 2017 operational classification of seizure types. Epilepsia. 2017 Apr;58(4):531-542. doi: 10.1111/epi.13671. Epub 2017 Mar 8. PMID 28276064
- [Background] Gaillard WD, Chiron C, Cross JH, Harvey AS, Kuzniecky R, Hertz-Pannier L, Vezina LG; ILAE, Committee for Neuroimaging, Subcommittee for Pediatric. Guidelines for imaging infants and children with recent-onset epilepsy. Epilepsia. 2009 Sep;50(9):2147-53. doi: 10.1111/j.1528-1167.2009.02075.x. Epub 2009 Apr 6. PMID 19389145
- [Background] D'Argenzio L, Colonnelli MC, Harrison S, Jacques TS, Harkness W, Vargha-Khadem F, Scott RC, Cross JH. Cognitive outcome after extratemporal epilepsy surgery in childhood. Epilepsia. 2011 Nov;52(11):1966-72. doi: 10.1111/j.1528-1167.2011.03272.x. PMID 22032791